CLINICAL TRIAL: NCT02821234
Title: The Sleepless Brain: Neuroimaging Support for a Differential Diagnosis of Insomnia
Acronym: SOMNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut des Maladies Neurodégénératives (UMR5293) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2016/05
Record Dates: First submitted 2016-06-17; First posted 2016-07-01 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Insomnia
Keywords: Insomnia; Hyperarousal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insomnia group (Experimental): Patients with insomnia: sleep complaints, of at least 3 nights a week, for at least 3 months, affected daytime functioning, objectified low sleep quality (SE <85%) with 10 days actigraphy occurred in the last 2 months
  Interventions: Other: MRI
- Control group (Experimental): Volunteer without sleep problems either self-reported or objectified through actigraphy (SE ≥85%)
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI

SUMMARY:
One-tenth of the population suffers from insomnia, increasing their risk on other health problems such as depression. Self-reported sleep quality only was historically leading for insomnia diagnosis, but more recently a state of 24-hour hyperarousal has been associated with insomnia, either physiological (increased heart rate, higher frequency EEG) or predominant cognitive-emotional hyperarousal (worry, rumination, repetitive thoughts). Strong evidence shows that those suffering from insomnia with physiological hyperarousal are at higher risk of short and long term severe health problems such as inflammation and hypertension than the group without physiological hyperarousal. The neurophysiological basis of these insomnia phenotypes has however barely been investigated, although its results can have major consequences for how this limiting condition will be treated.

To support the development of a differential diagnosis of insomnia, structural and functional brain connectivity in insomnia patients with different levels of hyperarousal will be investigated and related to sleep variables. Investigators will compare the insomnia group to a normal sleeping control group. Investigators expect that the emotion processing circuit (amygdala-ventromedial prefrontal cortex) is a) more affected in insomniacs compared to normal sleeping controls and b) the directionality of this effect to depend on the level and type of hyperarousal in insomniacs. Further, investigators expect c) amygdala activity to be positive correlated with physiological hyperarousal level and d) prefrontal activity to be positively correlated with cognitive-emotional hyperarousal level. Investigators expect a higher physiological hyperarousal level to be reflected in affected afferent pathways of the amygdala towards the ventromedial prefrontal cortex and investigators expect higher cognitive-emotional hyperarousal to be related to affected efferent pathways from the ventromedial prefrontal cortex to the amygdala. Investigators expect sleep quality to play a mediating role in both types of hyperarousal and their brain activation patterns in insomnia patients and normal sleeping controls.

These data can lead to the definition of new insomnia phenotypes and to new customized and effective insomnia treatment, focused not only on improving sleep but also on changing dysfunctional hyperarousal levels that currently put insomniacs at risk of numerous severe health problems.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia group: patients with insomnia: sleep complaints, of at least 3 nights a week, for at least 3 months, affected daytime functioning.
* control group: no self-reported sleep problems in the last 2 months.
* 20-50 years old.
* Male or female.
* having given written informed consent to participate in the research project.

Exclusion Criteria:

* Night and shift-workers.
* Psychiatric disorder: clinical mood disorder, anxiety disorder, psychosis, bipolar disorder.
* For insomnia group: all sleep disorders other than persistent insomnia.
* For control group: all sleep disorders.
* Progressive neurological diseases that include restless legs syndrome.
* Cardiovascular disease other than treated hypertension.
* Unstable respiratory or endocrinological diseases.
* Drug addiction, alcohol addiction during the previous 6 months.
* Having undertaken trans-meridian travel (± 3H) in the previous 1 month.
* Pregnant or lactating women.
* Chronic pain.
* Hypnotic and psychotropic medication taking or stopped less than 5 half-life periods of molecules before screening V0.
* Patient participating to any other interventional study.
* For MRI: presence of a ferromagnetic foreign body (in particular certain intracranial clips, certain cardiac valves, intraocular foreign body, or subject having worked with metals), the presence of an implanted pacemaker, subject with cardiac or brain valves of ventricular derivation (risk of maladjustment), claustrophobia.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Resting state intrinsic connectivity within the emotion processing network by MRI | During Visit V2 (study termination), up to 3 month after consent signature

SECONDARY OUTCOMES:
Total sleep time obtained by actimetry | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Sleep efficiency obtained by actimetry | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Wake after sleep onset obtained by actimetry | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Sleep latency obtained by actimetry | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Total sleep time obtained by sleep diary | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Sleep efficiency obtained by sleep diary | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Wake after sleep onset obtained by sleep diary | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
sleep latency obtained by sleep diary | During the 10 nights preceding Inclusion Visit (up to 1 month after consent signature)
Questionnaire regarding sleep problems : Pittsburgh Sleep Questionaire (PSQ) | During Pre-inclusion Visit, at consent signature
Questionnaire regarding sleep problems : Insomnia Severity Index (ISI) | During Pre-inclusion Visit, at consent signature
Questionnaire regarding depression : Beck Depression Inventory (BDI) | During Pre-inclusion Visit, at consent signature
Questionnaire regarding anxiety : Beck Anxiety Inventory (BAI) | During Pre-inclusion Visit, at consent signature
Questionnaire regarding arousal : Arousal Predisposition Scale (APS) | During Inclusion Visit, up to 1 month after consent signature
Questionnaire regarding sleep reactivity : Ford Insomnia Response to Stress Test (FIRST) | During Inclusion Visit, up to 1 month after consent signature
Questionnaire regarding presleep arousal state : Presleep State Arousal Scale (PSAS) | During Visit V2 (study termination), up to 3 month after consent signature
Questionaire regarding emotional state : Positive and Negative Affect Schedule (PANAS) | During Visit V2 (study termination), up to 3 month after consent signature

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanz-Arigita E, Daviaux Y, Joliot M, Dilharreguy B, Micoulaud-Franchi JA, Bioulac S, Taillard J, Philip P, Altena E. Brain reactivity to humorous films is affected by insomnia. Sleep. 2021 Sep 13;44(9):zsab081. doi: 10.1093/sleep/zsab081. PMID 33772591